CLINICAL TRIAL: NCT03667131
Title: Effect of Prophylactic Treatment With Enalapril Maleate on Arterial Stiffness in Rheumatoid Arthritis Patients.
Brief Title: Enalapril Maleate on Arterial Stiffness in Rheumatoid Arthritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Mónica VázquezdelMercadoEspinosa, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EEVA
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Rheumatoid Arthritis
Keywords: arterial stiffness; enalapril maleate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Enalapril; Angiotensin-Converting Enzyme Inhibitors

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, controlled, parallel groups clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, care provider, investigator and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enalapril Maleate (Experimental): Enalapril Maleate 5 mg every 12 hrs for 90 days.
  Interventions: Drug: Enalapril Maleate
- Placebo (Experimental): Substance that lacks in itself therapeutic action.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enalapril Maleate — Enalapril Maleate 5 mg tablet, every 12 hrs for 90 days.
  Other Names: Angiotensin converting enzyme inhibitor.
  Arms: Enalapril Maleate
Drug: Placebo — Placebo 5 mg tablet, every 12 hrs for 90 days.
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
This study evaluates the effect in artery stiffness of enalapril maleate in Rheumatoid Arthritis women patients. Half of participants will receive 5 mg enalapril maleate every 12 hrs, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Rheumatoid Arthritis (RA) is a chronic inflammatory systemic disease considered as an independent cardiovascular risk factor that is associated with cumulative inflammatory load with an elevation of circulating levels of cytokines, which mediate the mechanism of endothelial cells activation by increasing the angiotensin converting enzyme (ACE) function and generation of vasoconstriction. Enalapril maleate is a prodrug that is hydrolyzed by hepatic esterases in enalaprilat, which is a potent inhibitor of ACE. ACE inhibition decreases vascular systemic resistance and mean, diastolic and systolic blood pressures in several hypertensive states, independently of the mechanism, ACE inhibitors have a widespread clinic use for cardiovascular diseases. Therefore, the researchers considered that there could be an association between the use of enalapril and the decrease in arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified with RA according to the American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) 2010
* Patients treated in the outpatient service of the Rheumatology Service of the Hospital Civil de Guadalajara "Dr. Juan I Menchaca".
* Sign an Informed Consent Letter
* Under treatment with conventional Disease-Modifying Antirheumatic Drugs (DMARDS)

Exclusion Criteria:

* Patients with a previous diagnosis of diabetes mellitus, systemic hypertension, thyroid, kidney or liver disease
* History of acute myocardial infarction, cardiac arrhythmias, cerebral vascular event or heart failure
* Smoking active patients in the last 6 months
* Patients with a desire for close conception, pregnant or breastfeeding.
* Patients with blood pressure <90/60 mmHg
* Patients who do not accept to participate in the study
* Patients with a BMI greater than ≥40 Kg / m2
* Non-palpable carotid and femoral pulses
* Unstable psychological state

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
Change in Pulse Wave Velocity (PWV) | Baseline and 90 days
  This is a measure of arterial stiffness, or the rate at which pressure waves move down the vessel.

SECONDARY OUTCOMES:
Change in Cardio-Ankle Vascular Index | Baseline and 90 days
  This is calculated from PWV at the origin of the aorta to the ankle portion of the tibial artery, and systolic and diastolic blood pressures measured at the upper brachial artery.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Vázquez-Del Mercado, MD, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Investigación en Reumatología y Sistema Músculo Esquelético, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for pulse wave velocity will be available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within one year of study completion.
Access Criteria: Data access requests will be reviewed by an external independent Review Panel. Requests will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Gossec L, Dougados M, Dixon W. Patient-reported outcomes as end points in clinical trials in rheumatoid arthritis. RMD Open. 2015 Apr 2;1(1):e000019. doi: 10.1136/rmdopen-2014-000019. eCollection 2015. PMID 26509052
- [Background] Burmester GR, Feist E, Dorner T. Emerging cell and cytokine targets in rheumatoid arthritis. Nat Rev Rheumatol. 2014 Feb;10(2):77-88. doi: 10.1038/nrrheum.2013.168. Epub 2013 Nov 12. PMID 24217582
- [Background] Gibofsky A. Overview of epidemiology, pathophysiology, and diagnosis of rheumatoid arthritis. Am J Manag Care. 2012 Dec;18(13 Suppl):S295-302. PMID 23327517
- [Background] Gkaliagkousi E, Gavriilaki E, Doumas M, Petidis K, Aslanidis S, Stella D. Cardiovascular risk in rheumatoid arthritis: pathogenesis, diagnosis, and management. J Clin Rheumatol. 2012 Dec;18(8):422-30. doi: 10.1097/RHU.0b013e31827846b1. PMID 23188207
- [Background] Solomon DH, Karlson EW, Rimm EB, Cannuscio CC, Mandl LA, Manson JE, Stampfer MJ, Curhan GC. Cardiovascular morbidity and mortality in women diagnosed with rheumatoid arthritis. Circulation. 2003 Mar 11;107(9):1303-7. doi: 10.1161/01.cir.0000054612.26458.b2. PMID 12628952
- [Background] Kramer HR, Giles JT. Cardiovascular disease risk in rheumatoid arthritis: progress, debate, and opportunity. Arthritis Care Res (Hoboken). 2011 Apr;63(4):484-99. doi: 10.1002/acr.20386. No abstract available. PMID 21452262
- [Background] Crowson CS, Nicola PJ, Kremers HM, O'Fallon WM, Therneau TM, Jacobsen SJ, Roger VL, Ballman KV, Gabriel SE. How much of the increased incidence of heart failure in rheumatoid arthritis is attributable to traditional cardiovascular risk factors and ischemic heart disease? Arthritis Rheum. 2005 Oct;52(10):3039-44. doi: 10.1002/art.21349. PMID 16200583
- [Background] Kremers HM, Crowson CS, Therneau TM, Roger VL, Gabriel SE. High ten-year risk of cardiovascular disease in newly diagnosed rheumatoid arthritis patients: a population-based cohort study. Arthritis Rheum. 2008 Aug;58(8):2268-74. doi: 10.1002/art.23650. PMID 18668561
- [Background] Crilly MA, Kumar V, Clark HJ, Scott NW, Macdonald AG, Williams DJ. Arterial stiffness and cumulative inflammatory burden in rheumatoid arthritis: a dose-response relationship independent of established cardiovascular risk factors. Rheumatology (Oxford). 2009 Dec;48(12):1606-12. doi: 10.1093/rheumatology/kep305. Epub 2009 Oct 25. PMID 19858120
- [Background] Klocke R, Cockcroft JR, Taylor GJ, Hall IR, Blake DR. Arterial stiffness and central blood pressure, as determined by pulse wave analysis, in rheumatoid arthritis. Ann Rheum Dis. 2003 May;62(5):414-8. doi: 10.1136/ard.62.5.414. PMID 12695151
- [Background] Park S, Lakatta EG. Role of inflammation in the pathogenesis of arterial stiffness. Yonsei Med J. 2012 Mar;53(2):258-61. doi: 10.3349/ymj.2012.53.2.258. PMID 22318811
- [Background] Roman MJ, Devereux RB, Schwartz JE, Lockshin MD, Paget SA, Davis A, Crow MK, Sammaritano L, Levine DM, Shankar BA, Moeller E, Salmon JE. Arterial stiffness in chronic inflammatory diseases. Hypertension. 2005 Jul;46(1):194-9. doi: 10.1161/01.HYP.0000168055.89955.db. Epub 2005 May 23. PMID 15911740
- [Background] Vazquez-Del Mercado M, Nunez-Atahualpa L, Figueroa-Sanchez M, Gomez-Banuelos E, Rocha-Munoz AD, Martin-Marquez BT, Corona-Sanchez EG, Martinez-Garcia EA, Macias-Reyes H, Gonzalez-Lopez L, Gamez-Nava JI, Navarro-Hernandez RE, Nunez-Atahualpa MA, Andrade-Garduno J. Serum levels of anticyclic citrullinated peptide antibodies, interleukin-6, tumor necrosis factor-alpha, and C-reactive protein are associated with increased carotid intima-media thickness: a cross-sectional analysis of a cohort of rheumatoid arthritis patients without cardiovascular risk factors. Biomed Res Int. 2015;2015:342649. doi: 10.1155/2015/342649. Epub 2015 Mar 2. PMID 25821796
- [Background] Wallberg-Jonsson S, Caidahl K, Klintland N, Nyberg G, Rantapaa-Dahlqvist S. Increased arterial stiffness and indication of endothelial dysfunction in long-standing rheumatoid arthritis. Scand J Rheumatol. 2008 Jan-Feb;37(1):1-5. doi: 10.1080/03009740701633238. PMID 18189187
- [Background] Vazquez-Del Mercado M, Gomez-Banuelos E, Chavarria-Avila E, Cardona-Munoz E, Ramos-Becerra C, Alanis-Sanchez A, Cardona-Muller D, Grover-Paez F, Perez-Vazquez FJ, Navarro-Hernandez RE, Valadez-Soto JM, Saldana-Millan AA, Gonzalez-Rosas L, Ramos-Lopez G, Petri MH, Back M. Disease duration of rheumatoid arthritis is a predictor of vascular stiffness: a cross-sectional study in patients without known cardiovascular comorbidities: A STROBE-compliant article. Medicine (Baltimore). 2017 Aug;96(33):e7862. doi: 10.1097/MD.0000000000007862. PMID 28816989
- [Derived] Perez-Vazquez F, Back M, Chavarria-Avila E, Gomez-Banuelos E, Ramos-Becerra CG, Pizano-Martinez O, Salazar-Paramo M, Grover-Paez F, Nava-Zavala AH, Cardona-Munoz EG, Cardona-Muller D, Duran-Barragan S, Mera-Riofrio VN, Prado-Bachega N, Vazquez-Del Mercado M. Enalapril Influence on Arterial Stiffness in Rheumatoid Arthritis Women: A Randomized Clinical Trial. Front Med (Lausanne). 2020 Jan 29;6:341. doi: 10.3389/fmed.2019.00341. eCollection 2019. PMID 32118001